CLINICAL TRIAL: NCT06281301
Title: Improving Patient Understanding of Macrosomia: a Randomized Control Trial
Brief Title: Improving Patient Understanding of Macrosomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kristen Cagino, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-23-1023
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Macrosomia, Fetal
MeSH Terms: conditions — Fetal Macrosomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no additional information (Other)
  Interventions: Other: no additional information
- education tool (Experimental)
  Interventions: Other: education tool

INTERVENTIONS:
Other: education tool — Participants will have 15 minutes to review the single sided card and then the survey will be administered. Participants will then be surveyed again within 1-2 weeks after initial completion to assess how well information was retained.
  Arms: education tool
Other: no additional information — Survey will be administered without reviewing the single sided card
  Arms: no additional information

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a graphic based education tool on patient knowledge of macrosomia through the use of a survey and to evaluate knowledge at 1-2 weeks after initial review of the education tool.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* greater than or equal to 36 weeks gestation.

Exclusion Criteria:

* unable to provide informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Number of participants that showed Macrosomia knowledge as assessed by the score on a survey | immediately after intervention (about 5 minutes after intervention)
  This survey has 17 questions and will be scored from 1-17 higher number indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Cagino, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No